CLINICAL TRIAL: NCT00130832
Title: Safety and Immunogenicity of Concomitant Use and Staggered Use of Vaccine and Oral Poliovirus (OPV) in Healthy Infants
Brief Title: Concomitant Use and Staggered Use of Vaccine and Oral Poliovirus (OPV) in Healthy Infants (V260-014)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V260-014; 2005_030
Record Dates: First submitted 2005-08-12; First posted 2005-08-16 (Estimated); Results first posted 2010-09-09 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Rotavirus Infections; Gastroenteritis
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis | interventions — Rotavirus Vaccines; Poliovirus Vaccine, Oral

ARMS (2):
- 1 (Experimental): RotaTeq and OPV concomitantly
  Interventions: Biological: Rotavirus Vaccine, Live, Oral, Pentavalent; Biological: Comparator: Oral Poliovirus Vaccine (OPV)
- 2 (Experimental): RotaTeq and OPV on staggered schedule
  Interventions: Biological: Rotavirus Vaccine, Live, Oral, Pentavalent; Biological: Comparator: Oral Poliovirus Vaccine (OPV) (staggered)

INTERVENTIONS:
Biological: Rotavirus Vaccine, Live, Oral, Pentavalent — Three doses of rotavirus vaccine, live, oral, pentavalent. Dose 1 was given on Day 1, Dose 2 was given 56 to 84 days post Dose 1, and Dose 3 was given 56 to 84 days post Dose 2.
Biological: Comparator: Oral Poliovirus Vaccine (OPV) — Three doses OPV. Dose 1 was given on Day 1, Dose 2 was given 56 to 84 days post Dose 1, and Dose 3 was given 56 to 84 days post Dose 2.
  Arms: 1
Biological: Comparator: Oral Poliovirus Vaccine (OPV) (staggered) — Three doses OPV. Dose 1 was given 14 to 28 days post Dose 1 of RotaTeq, Dose 2 was given 14 to 28 days post Dose 2 of RotaTeq, and Dose 3 was given 14 to 28 days post Dose 3 of RotaTeq.
  Arms: 2

SUMMARY:
The study is being conducted to demonstrate that vaccine to prevent gastroenteritis due to rotavirus may be administered concomitantly with oral polio vaccine (OPV) without impairing the safety or immunogenicity of either vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Infants in good health

Exclusion Criteria:

* Previous administration of any oral poliovirus vaccine (OPV) and rotavirus vaccine
* Receipt of inactivated poliovirus vaccine (IPV) prior to the first dose of either study vaccine, or at any time during the course of the study
* Any condition resulting in depressed immunity
* Any allergy to any vaccine component as stated in the package circulars
* Allergies to polymyxin B, neomycin or any other antibiotics
* Receipt of intramuscular, oral, or intravenous corticosteroid treatment
* History of congenital abdominal disorders, intussusception, or abdominal surgery; clinical evidence of active gastrointestinal illness
* History of known prior rotavirus gastroenteritis, chronic diarrhea, or failure to thrive
* Prior receipt of a blood transfusion or blood products, including immunoglobulin
* Fever, with a rectal temperature of ≥38.1°C (≥ 100.5°F) at the time of immunization
* Infants residing in a household with an immunocompromised person

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 735 (Actual)
Dates: Start 2005-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Ciarlet M, Sani-Grosso R, Yuan G, Liu GF, Heaton PM, Gottesdiener KM, Arredondo JL, Schodel F. Concomitant use of the oral pentavalent human-bovine reassortant rotavirus vaccine and oral poliovirus vaccine. Pediatr Infect Dis J. 2008 Oct;27(10):874-80. doi: 10.1097/INF.0b013e3181782780. PMID 18756184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred at 9 study sites in Mexico, Costa Rica, Guatemala, and Brazil from 19-Oct-2005 (first subject in) to 06-Jan-2006 (last subject randomized).
Pre-assignment Details: Excluded from randomization were subjects with history of congenital abdominal disorders, intussusception, or abdominal surgery; history of known prior rotavirus disease, chronic diarrhea, or failure to thrive, clinical evidence of active gastrointestinal illness and those with fever, a rectal temperature ≥38.1°C (≥100.5°F) at time of immunization.
Groups:
- RotaTeq and Oral Poliovirus (OPV) Concomitantly: Subjects (Sbjs) in Group 1 who received 3 concomitant doses of RotaTeq™ and OPV ≥56 to ≤84 days (8 to 10 weeks) apart
- RotaTeq and Oral Poliovirus (OPV) Staggered: Subjects in Group 2, who received RotaTeq™ first followed by OPV between ≥14 to ≤28 days (2 to 4 weeks) later
Period: Overall Study
Arm/Group | RotaTeq and Oral Poliovirus (OPV) Concomitantly | RotaTeq and Oral Poliovirus (OPV) Staggered
Started | 372 | 363
Completed | 356 (Those who received all 3 doses of concomitant RotaTeq™/ OPV with blood draw ~42 days postdose 3) | 346 (Those who received all 3 doses; last 2 blood draws ~42 days postdose 3 of RotaTeq™ and postdose OPV)
Not Completed | 16 | 17
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 6 | 8
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Moved | 2 | 2
Not completed — Other | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RotaTeq and Oral Poliovirus (OPV) Concomitantly | RotaTeq and Oral Poliovirus (OPV) Staggered | Total
Number analyzed (Participants) | 372 | 363 | 735
Age, Customized [Number; unit: participants]
  5 Weeks of Age and Under | 8 | 1 | 9
  6 to 12 Weeks of Age | 364 | 362 | 726
  Over 12 Weeks of Age | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 194 | 383
  Male | 183 | 169 | 352
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2 | 1 | 3
  Black | 10 | 7 | 17
  Hispanic American | 263 | 257 | 520
  Multi-Racial | 56 | 61 | 117
  White | 41 | 37 | 78

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer(s) of Poliovirus Types 1, 2, and 3, Measured Approximately 42 Days Postdose 3
Description: GMT of poliovirus type 1, 2, and 3, measured at postdose 3 in subjects receiving RotaTeq™ and OPV concomitantly compared to staggered.
Time Frame: Approximately 42 days Postdose 3
Population: The primary immunogenicity analyses were based on evaluable per-protocol subjects who received all scheduled doses, were not protocol violators, and had valid assay values.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titer (GMT)
Arm/Group | RotaTeq and Oral Poliovirus (OPV) Concomitantly | RotaTeq and Oral Poliovirus (OPV) Staggered
Number analyzed (Participants) | 355 | 318
Geometric Mean Titer (GMT)
  Antibody Responses to Poliovirus Type 1 | 888.0 [752.8 to 1047] | 1139 [969.1 to 1340]
  Antibody Responses to Poliovirus Type 2 | 814.9 [720.7 to 921.4] | 814.5 [707.4 to 937.9]
  Antibody Responses to Poliovirus Type 3 | 233.6 [201.9 to 270.2] | 269.2 [230.6 to 314.2]
Statistical Analysis 1: Comparison: RotaTeq and Oral Poliovirus (OPV) Concomitantly vs RotaTeq and Oral Poliovirus (OPV) Staggered; Seroprotection rate (proportion of subjects who achieve the seroprotection criteria: neutralizing antibody titers [NA] ≥1:8) for poliovirus type 1; Test type: Non-Inferiority or Equivalence — non-inferiority criterion is that the lower limit of the 2-sided 95% confidence interval of the proportion difference (concomitant group minus staggered group) for subjects who achieve neutralizing antibody titers [NA] ≥1:8 greater than -10%; p < 0.001, Miettinen and Nurminen's; Comparing seroprotection rate difference with the non-inferiority margin of 0.10 with Miettinen and Nurminen's method; Seroprotection Rate Difference = -0.5, 95% CI [-2.2 to 1.4]
Statistical Analysis 2: Comparison: RotaTeq and Oral Poliovirus (OPV) Concomitantly vs RotaTeq and Oral Poliovirus (OPV) Staggered; Seroprotection rate (proportion of subjects who achieve the seroprotection criteria: neutralizing antibody titers [NA] ≥1:8) for poliovirus type 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen's; Comparing seroprotection rate difference with the non-inferiority margin of 0.10 with Miettinen and Nurminen's method; Seroprotection Rate Difference = 0.0, 95% CI [-1.4 to 1.6]
Statistical Analysis 3: Comparison: RotaTeq and Oral Poliovirus (OPV) Concomitantly vs RotaTeq and Oral Poliovirus (OPV) Staggered; Seroprotection rate (proportion of subjects who achieve the seroprotection criteria: neutralizing antibody titers [NA] ≥1:8) for poliovirus type 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen's; Comparing seroprotection rate difference with the non-inferiority margin of 0.10 with Miettinen and Nurminen's method; Seroprotection Rate Difference = -0.1, 95% CI [-2.3 to 2.3]

2. Primary Outcome: GMT of Serum Anti-rotavirus Immunoglobulin A (IgA)
Description: GMT of serum anti-rotavirus IgA measured at postdose 3 in subjects receiving RotaTeq™ and OPV concomitantly compared to staggered
Time Frame: Approximately 42 days Postdose 3
Population: Per Protocol Population
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | RotaTeq and Oral Poliovirus (OPV) Concomitantly | RotaTeq and Oral Poliovirus (OPV) Staggered
Number analyzed (Participants) | 351 | 320
GMT | 154.9 [126.4 to 189.9] | 292.7 [248.6 to 344.6]
Statistical Analysis 1: Comparison: RotaTeq and Oral Poliovirus (OPV) Concomitantly vs RotaTeq and Oral Poliovirus (OPV) Staggered; Test type: Non-Inferiority or Equivalence — non-inferiority criterion is that the lower limit of the 2-sided 95% confidence interval of the GMT ratio (concomitant group over staggered group) greater than 0.50; p = 0.277, ANOVA; ANOVA model on log titer of serum anti-rotavirus IgA; GMT Ratio = 0.54, 95% CI [0.42 to 0.69]
Statistical Analysis 2: Comparison: RotaTeq and Oral Poliovirus (OPV) Concomitantly vs RotaTeq and Oral Poliovirus (OPV) Staggered; Test type: Non-Inferiority or Equivalence — non-inferiority criterion is that the lower limit of the 2-sided 95% confidence interval of the proportion difference (concomitant group minus staggered group) for subjects who achieve 3-fold rise in serum anti-rotavirus IgA greater than -10%; p = 0.002, Miettinen and Nurminen's; Comparing percentage difference with the non-inferiority margin of 10 percentage point with Miettinen and Nurminen's method; Percentage Point Difference = -4.4, 95% CI [-8.0 to -1.4] — Percentage point difference (concomitant - staggered)

3. Primary Outcome: Immunogenicity of RotaTeq™ as Measured by Serum Neutralizing Antibody [SNA] Responses to Rotavirus Serotypes G1, G2, G3, G4, and P1A When Administered With OPV Concomitantly or Staggered
Description: Rotavirus SNA response to serotypes G1, G2, G3, G4, and P1A measured at postdose 3 in subjects receiving RotaTeq™ and OPV concomitantly compared to staggered.
Time Frame: Approximately 42 days Postdose 3
Population: Per Protocol Population
  For serotype G4 the RotaTeq and Oral Poliovirus (OPV) concomitantly group N = 350
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | RotaTeq and Oral Poliovirus (OPV) Concomitantly | RotaTeq and Oral Poliovirus (OPV) Staggered
Number analyzed (Participants) | 352 | 321
GMT
  SNA responses to rotavirus serotypes G1 | 125.8 [106.7 to 148.2] | 182.6 [158.2 to 210.7]
  SNA responses to rotavirus serotypes G2 | 27.1 [22.9 to 32.0] | 30.0 [25.9 to 34.8]
  SNA responses to rotavirus serotypes G3 | 21.2 [18.4 to 24.32] | 22.5 [19.4 to 26.0]
  SNA responses to rotavirus serotypes G4 | 58.5 [50.2 to 68.1] | 74.5 [64.3 to 86.3]
  SNA responses to rotavirus serotypes P1A | 84.7 [71.97 to 99.8] | 131.4 [112.6 to 153.2]

ADVERSE EVENTS:
Time Frame: Subjects in this study were followed for all adverse experiences, for 14 days following each study vaccination.
Description: The number of subjects listed in the Adverse Event tables is the number of subjects who received study treatment.
  Although a subject may have had two or more clinical adverse experiences the patient is counted only once in a category. The same subject may appear in different categories.
Arm/Group | RotaTeq and Oral Poliovirus (OPV) Concomitantly | RotaTeq and Oral Poliovirus (OPV) Staggered
Serious Adverse Events (participants affected / at risk) | 4/366 | 9/359
Other Adverse Events (participants affected / at risk) | 342/366 | 325/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RotaTeq and Oral Poliovirus (OPV) Concomitantly (N=366) | RotaTeq and Oral Poliovirus (OPV) Staggered (N=359)
Intussusception (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Bronchiolitis (Infections and infestations) | 2 | 0
Meningitis pneumococcal (Infections and infestations) | 1 | 0
Pertussis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RotaTeq and Oral Poliovirus (OPV) Concomitantly (N=366) | RotaTeq and Oral Poliovirus (OPV) Staggered (N=359)
Conjunctivitis (Eye disorders) | 8 | 7
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Constipation (Gastrointestinal disorders) | 13 | 18
Diarrhoea (Gastrointestinal disorders) | 195 | 185
Flatulence (Gastrointestinal disorders) | 7 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 5
Infantile colic (Gastrointestinal disorders) | 34 | 37
Vomiting (Gastrointestinal disorders) | 123 | 121
Influenza like illness (General disorders) | 7 | 8
Injection site pain (General disorders) | 16 | 21
Irritability (General disorders) | 24 | 33
Pain (General disorders) | 3 | 6
Pyrexia (General disorders) | 203 | 202
Bronchiolitis (Infections and infestations) | 10 | 9
Bronchitis (Infections and infestations) | 5 | 4
Ear infection (Infections and infestations) | 6 | 5
Influenza (Infections and infestations) | 28 | 38
Nasopharyngitis (Infections and infestations) | 85 | 86
Oral candidiasis (Infections and infestations) | 7 | 4
Otitis media (Infections and infestations) | 2 | 5
Pharyngitis (Infections and infestations) | 32 | 37
Rhinitis (Infections and infestations) | 14 | 17
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 18
Headache (Nervous system disorders) | 2 | 4
Crying (Psychiatric disorders) | 3 | 5
Restlessness (Psychiatric disorders) | 8 | 16
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 54 | 52
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 16 | 19
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Dermatitis (Skin and subcutaneous tissue disorders) | 9 | 13
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 8 | 5
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 11 | 9
Rash (Skin and subcutaneous tissue disorders) | 5 | 7
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.